CLINICAL TRIAL: NCT00115453
Title: Boron Neutron Capture Therapy in the Treatment of Glioblastoma Multiforme
Brief Title: Boron Neutron Capture Therapy (BNCT) as Treatment of Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Boneca Corporation (Industry)
Responsible Party: CEO Markku Pohjola, BONECA Ltd, Tukholmankatu 8
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNCT-P01
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Glioblastoma
Keywords: glioblastoma; boron neutron capture therapy; boronophenylalanine; brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Active treatment arm.
  Interventions: Radiation: irradiation

INTERVENTIONS:
Radiation: irradiation — Boronophenylalanine is infused into a peripheral vein prior to neutron irradiation.

SUMMARY:
Boron Neutron Capture Therapy (BNCT) is an experimental radiation therapy technique that is based on the principle of irradiating boron atoms with neutrons. When neutrons have relatively low energy, boron atoms that have been targeted to cancerous tissue using a suitable boron carrier (an amino acid derivative called BPA, boronophenylalanine) will capture the neutrons. As a result from the neutron capture the boron atoms will split into two, producing helium and lithium ions. The helium and lithium ions, in turn, have only a short pathlength in tissue (about 5 micrometers) and will deposit their cell damaging effect mainly within the tumor provided that the boron carrier (BPA) has accumulated in the tumor. In practice, the study participants will receive BPA as an approximately 2-hour intravenous infusion, following which the tumor is irradiated with low energy (epithermal) neutrons obtained from a nuclear reactor at the BNCT facility. BNCT requires careful radiation dose planning, but neutron irradiation will last approximately only for one hour. In this study BNCT is given only once. The study hypothesis is that glioblastoma tissue may accumulate the boron carrier compound, and glioblastoma might respond to BNCT.

DETAILED DESCRIPTION:
This is a single BNCT-facility, non-randomized, non-comparative, prospective, open-label, phase I/II trial to determine the value of BNCT in the treatment of subjects who have undergone surgery for glioblastoma, but glioblastoma has not been treated with radiation therapy or chemotherapy. The neutron irradiation site is the FiR 1 reactor site, located at Otaniemi, Espoo, Finland, about 6 kilometers from the Helsinki University Central Hospital, Helsinki, where patient evaluation and post-irradiation care will take place.

BPA is infused as a fructose complex (BPA-F) into a peripheral vein over 2 hours prior to neutron irradiation. Blood samples will be taken before starting the BPA infusion, and thereafter at 20 to 40 minute intervals during the infusion, following infusion, and after delivering neutron irradiation to monitor the blood boron concentration. The blood samples will be analyzed for boron to estimate the average blood boron level during neutron irradiation. The first 12 patients are treated using a BPA dose of 290 mg/kg, following which the dose of BPA is increased stepwise to 500 mg/kg, provided that unacceptable toxicity will not occur.

All patients will be evaluated for response using CT or magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme
* Supratentorial location
* At least 30% of the tumor volume has been removed at craniotomy as judged from a pre/perioperative MRI
* Ability to understand the concept of investigational therapy
* Tolerates dexamethasone treatment
* Adequate anti-epileptic medication
* BNCT can be delivered within 6 weeks from the date of brain surgery
* A written informed consent

Exclusion Criteria:

* Age less than 18 or greater than 75
* The tumor infiltrates into the optic chiasm or into the deep parts of the brain prohibiting delivery of an adequate radiation dose with BNCT
* Prior radiation therapy to the brain
* Prior chemotherapy, immunotherapy, or gene therapy
* Karnofsky performance score <70
* Severe cardiac, liver, or kidney failure
* Severe infection
* A cardiac pace-maker, or a metal implant in the head and neck region that will prohibit MRI examination
* Pregnancy or lactation
* Phenylketonuria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1999-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
safety | 3 years

SECONDARY OUTCOMES:
tumor response | one year
effect on brain tissue | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, M.D., prof., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Kouri M, Kankaanranta L, Seppala T, Tervo L, Rasilainen M, Minn H, Eskola O, Vahatalo J, Paetau A, Savolainen S, Auterinen I, Jaaskelainen J, Joensuu H. Undifferentiated sinonasal carcinoma may respond to single-fraction boron neutron capture therapy. Radiother Oncol. 2004 Jul;72(1):83-5. doi: 10.1016/j.radonc.2004.03.016. PMID 15236879
- [Result] Joensuu H, Kankaanranta L, Seppala T, Auterinen I, Kallio M, Kulvik M, Laakso J, Vahatalo J, Kortesniemi M, Kotiluoto P, Seren T, Karila J, Brander A, Jarviluoma E, Ryynanen P, Paetau A, Ruokonen I, Minn H, Tenhunen M, Jaaskelainen J, Farkkila M, Savolainen S. Boron neutron capture therapy of brain tumors: clinical trials at the finnish facility using boronophenylalanine. J Neurooncol. 2003 Mar-Apr;62(1-2):123-34. doi: 10.1007/BF02699939. PMID 12749708